CLINICAL TRIAL: NCT06425965
Title: Effect of Hybrid Simulation Method on Advanced Life Support Application of Nursing Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yagmur Sen, Research Assistant, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 641752
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Advanced Life Support; Simulation Training; Nursing Education
Keywords: simulation; Advanced life support; Nursing education; Nursing student; Web-based simulation; High fadility

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group 1 (Experimental): The first group will receive advanced life support training with a high reality simulator.
  Interventions: Other: Advanced life support training with high reality simulator
- Intervention Group 2 (Experimental): The second group will receive advanced life support training with web-based simulation method.
  Interventions: Other: Advanced life support training with web-based simulation
- Intervention Group 3 (Experimental): The third group will receive advanced life support training with a hybrid simulation method using both high reality simulator and web-based simulation.
  Interventions: Other: Advanced life support training with hybrid simulation

INTERVENTIONS:
Other: Advanced life support training with high reality simulator — The training consists of theoretical and practical training and lasts 3 hours a day, 5 days, for a total of 15 hours. The first 3 days of the training are theoretical, 1 day is laboratory practice and 1 day is evaluation. Theoretical courses start with introductions and sharing the content of the training and aim to provide the basic professional knowledge and skills required for advanced life support practice (diagnosis of cardiac arrest, ensuring airway patency, monitoring, cardiac rhythm diagnosis, drugs used during advanced life support and advanced life support algorithm). The laboratory application of the training is carried out with a high reality simulator in line with the information (15 min), scenario implementation (15 min) and debriefing sessions (30 min), respectively.
  Arms: Intervention Group 1
Other: Advanced life support training with web-based simulation — The training consists of theoretical and practical training and lasts 3 hours a day, 5 days, for a total of 15 hours. The first 3 days of the training are theoretical, 1 day is laboratory practice and 1 day is evaluation. Theoretical courses start with introductions and sharing the content of the training and aim to provide the basic professional knowledge and skills required for advanced life support practice (diagnosis of cardiac arrest, ensuring airway patency, monitoring, cardiac rhythm diagnosis, drugs used during advanced life support and advanced life support algorithm). The laboratory application of the training is carried out by web-based simulation method. Students participate in the web-based simulation application developed by the researcher.
  Arms: Intervention Group 2
Other: Advanced life support training with hybrid simulation — The training consists of theoretical and practical training and lasts 3 hours a day, 5 days, for a total of 15 hours. The first 3 days of the training are theoretical, 1 day is laboratory practice and 1 day is evaluation. Theoretical courses start with introductions and sharing the content of the training and aim to provide the basic professional knowledge and skills required for advanced life support practice (diagnosis of cardiac arrest, ensuring airway patency, monitoring, cardiac rhythm diagnosis, drugs used during advanced life support and advanced life support algorithm). The laboratory application of the training is carried out with the hybrid simulation method in which high reality simulator and web-based simulation method are applied together. Students first apply the web-based simulation developed by the researcher. Then they perform the practice on the high reality simulator.
  Arms: Intervention Group 3

SUMMARY:
The use of simulation in nursing education is an effective way to provide professional skills and enrich learning experiences while protecting patient safety. When the literature is examined, it is seen that simulation is frequently used in advanced life support training. The aim of the study is to examine the effects of advanced life support training in adults, which will be carried out with high-reality simulator/model simulation, web-based simulation and hybrid simulation methods, on the knowledge and skills of nursing students. It has been determined that training provided with hybrid simulation contributes to the professional development of students by creating individualized and interactive learning environments, and that students can more easily transfer the knowledge they have acquired in the educational environment to clinical practice. As a hybrid simulation method in the study; It is planned to use a combination of high-reality simulator/model, which has been proven to be effective in the development of psychomotor skills, and the web-based simulation method, which is effective in creating permanent learning by allowing students to repeat more. In the literature; It has been stated that the level of knowledge and skills gradually decreases after 6-10 weeks of advanced/basic life training. It is anticipated that the web-based simulation method will be effective in providing permanent learning as it gives learners the opportunity to repeat during/after the training. Based on these assumptions, it is planned to develop an adult advanced life support training program consisting of theory and practice, in which the development of students' professional skills is supported through hybrid simulation applications, and the students are provided with the opportunity to repeat. Since the study tests 3 different interventions, it is anticipated that it will lay the groundwork for subsequent studies and provide comprehensive information about simulation-based education practices.

ELIGIBILITY:
Inclusion Criteria:

* To complete first aid, internal medicine nursing, surgical nursing courses,
* Volunteering to participate in the research.
* Having experienced the simulation application before

Exclusion Criteria:

* Fail the specified courses (taking FF)
* Not having taken first aid course/training before
* Not having experienced the simulation application before.

Disqualification criteria:

* Being absent for more than 20% of the theoretical part of the planned advanced life support training
* Not participating in the laboratory applications of the planned advanced life support training
* Not having completed the planned web-based simulation application

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Advanced Life Support Knowledge Test | before training, immediately after training, 1 month after training, 3 months after training
  It was developed by the researchers in line with the literature to determine the level of knowledge of the participants about advanced life support practice.
Advanced Life Support Skill Checklist | before training, immediately after training, 1 month after training, 3 months after training
  It was developed by the researcher based on the European Resuscitation Council 2021 Advanced Life Support Algorithm.

SECONDARY OUTCOMES:
Student Satisfaction and Self-confidence in Learning Scale | immediately after training
  The scale was developed by Jeffries and Rizzolo in 2006. The Turkish validity and reliability study of the scale was conducted by Ünver et al. in 2015. The scale aims to determine students' satisfaction and self-confidence towards learning in simulation environment. The scale consists of two sub-dimensions, "Satisfaction with Current Learning" and "Confidence in Learning", and a total of 12 items. The scale is a 5-point Likert scale (1: Strongly disagree, 2: Disagree, 3: Undecided, 4: Agree, 5: Strongly Agree) and each item is scored as 1 being the lowest and 5 being the highest. The higher the total score obtained from the scale, the higher the student satisfaction and self-confidence in learning.
Simulation Design Scale | immediately after training
  The scale was developed by Jeffries and Rizzolo in 2006 and the Turkish validity and reliability study was conducted by Ünver et al. in 2015. The scale consists of 20 items and 2 sections. The first part measures simulation design elements, and the second part measures how important the simulation application is for students. An increase in the total score obtained in the first part of the scale indicates that the best simulation design elements are applied in the simulation application; an increase in the total score obtained from the second part indicates that the importance given by the student to the simulation experience is high.
Semi-structured Interview Form | immediately after training
  In this study, a semi-structured interview form developed by the researchers in line with the literature was used to determine the opinions of the students participating in the Advanced Life Support in Adults Training Program about the training program. The form consists of questions aimed at determining the theoretical content of the training program, the effectiveness of teaching methods (web-based simulation, simulation with high reality simulator, hybrid simulation), the effects of the training on learning retention, and suggestions for improving the training program.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Florence Nightingale Faculty of Nursing, Istanbul, Şişli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol